CLINICAL TRIAL: NCT05072561
Title: Feasibility of Radioisotope-guided Excision of Mediastinal Lymph Nodes in Patients With Non-small Cells Lung Carcinoma
Acronym: SLN_NSCLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1957
Record Dates: First submitted 2021-05-24; First posted 2021-10-11 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Diagnostic Test: Sentinel lymph node scintigraphy

INTERVENTIONS:
Diagnostic Test: Sentinel lymph node scintigraphy — During the surgery, right after the identification of the primary, 18-37 MBq of 99mTc-Nanocolloids in two ml will be injected at four peritumoral locations. After a brief waiting time (5-10'), the thoracic surgeon will perform the clinical intervention, including the lobectomy (the injection sites will be resected alongside the tumour) and lymphadenectomy, according to the best clinical practice. All the excised lymph nodes will be ex vivo counted using a gamma probe: those with a detectable activity (at least 10% of the "hottest" lymph node) will be considered as SLN. Thereafter, the mediastinum will be scanned using the gamma probe and a handheld gamma-camera (the latter will not be employed in case of robotic-assisted surgery); any further source of radioactivity will be investigated and, should further lymph nodes be identified, these will be also resected and classified in SLN or non-SLN, based on ex vivo activity.

SUMMARY:
Non-small cells lung carcinoma (NSCLC) represents one of the most common and lethal neoplasms. NSCLC is characterized by an early asymptomatic phase, which hinders the disease identification in its earliest stages. As a consequence, NSCLC is often diagnosed at a clinical stage when the potentially curative surgical approach is challenging. In general, NSCLC up to the TNM stage cT3N2M0 are considered operable; in particular, nodal localizations in the homolateral hilus (N1) and underneath the carina (N2) are considered surgically manageable. Identification of nodal disease on the pre-operative PET/CT does not guarantee that all disease-bearing lymph node will be retrieved in the course of the open operative procedure. Smaller nodes might be challenging to identify; moreover, the co-existence of macroscopic and microscopic disease might hinder the radicality of the surgical intervention. This process can be tracked using specific radioactive radiopharmaceuticals, such as radioisotope-labelled colloids, which can be injected in the immediate proximity of the primary and then travel toward the closest cluster of mediastinal lymph nodes. There, they are incorporated in the nodal structure and progress no farther. By employing a radioisotope probe during surgery, all of the first-line nodes (so-called sentinel lymph node, SLN), which receive the lymphatic flow from the tumor region directly, can be identified.

The hypothesis of the investigators is that, by performing a radioisotope SLN mapping intraoperatively, the surgeons will be able to detect the metastatization process more accurately than relying on pre-operative imaging alone.

The present study will be a prospective and monocentric trial. Clinical, histological, and imaging data collected from examinations performed according to the good clinical practice will be analyzed. The estimated duration of the study is 12 months. It will include the prospective inclusion of patients with a diagnosis of operable NSCLC, who will receive a surgical treatment with curative intent at the investigators' institution (ICH).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Newly diagnosis of stage I-IIIa NSCLC (higher stage could be considered, pending a multidisciplinary evaluation and approval).
* Baseline 18FFDG-PET-CT and ceCT
* Treatment according to good clinical practice

Exclusion criteria:

* Unavailability of baseline images
* Diagnosis other than NSCLC at definitive pathology
* Surgery carried without complete resection or with no curative intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Detection rate (DR) of the SLN technique. | 12 months
  The DR is defined as the capability of the SLN of identifying the mediastinal lymph nodes receiving the lymphatic flow, i.e., the presence and the number of lymph nodes, which can be identified with the gamma probe intraoperatively. This parameter will be measured as the ratio between the number of removed lymph nodes that will show a signifcant uptake of the radiotracer (>10 counts per minute) and the total number of removed lymph nodes.
Sensitivity (Se) of the SLN technique. | 12 months
  The Se will be defined as the ratio between the number of identified nodal disease foci that will show a signifcant uptake of the radiotracer (>10 counts per minute) and the total number of identified nodal disease foci.

SECONDARY OUTCOMES:
Measurement of the efficiency of a portable gamma camera | 12 months
  the measurement of the efficiency of a portable gamma camera, when compared with the standard gamma probe, in terms of DR. This parameter will be measured as the ratio between the number of removed lymph nodes that will show a signifcant uptake at the examination with the portable gamma camera (as evaluated by an expert operator) and the number of removed lymph nodes that will show a signifcant uptake of the radiotracer (>10 counts per minute) with the standard gamma probe
Comparison between the lower (I-II) and the higher (III and above) disease stages | 12 months
  The comparison of DR and Se between the lower (I-II) and the higher (III and above) disease stages. The analysis will be performed using the ROC curves for these parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No